CLINICAL TRIAL: NCT02176889
Title: A Double-blind, Placebo-controlled, Parallel Study Evaluating the Safety of Lactospore® in Healthy Individuals
Brief Title: A Parallel Study Evaluating the Safety of Lactospore® in Healthy Individuals
Acronym: 14PSHS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Sabinsa Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 14PSHS
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Lactospore; Bacillus coagulans; Safety; Probiotic; Healthy Adults; Tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactospore (Experimental): One tablet once daily, 30 minutes before a meal, preferably in the morning for 30 days
  Interventions: Dietary Supplement: Lactospore
- Placebo (Placebo Comparator): One tablet once daily, 30 minutes before a meal, preferably in the morning, for 30 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactospore — Bacillus coagulans MTCC 5856
  Arms: Lactospore
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Lactospore is safe in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* If female, subject is not of child bearing potential or female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
* Healthy as determined by laboratory results and medical history
* Normal BMI 18.5 - 29.9 kg/m2
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Subject has any clinically significant medical conditions
* Subject requires the use of prescribed medications (other than birth control)
* Use of illicit drugs or history of drug or alcohol abuse with the past 5 years (currently having more than 2 standard alcoholic drinks per day)
* Participation in a clinical research trial within 30 days prior to randomization
* Clinically significant abnormal laboratory results at screening
* Allergy or sensitivity to test product ingredients
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Lab parameters | Over 30 days
  CBC, electrolytes (Na, K, Cl), glucose, creatinine, AST, ALT, GGT, and bilirubin levels
Safety and Tolerability: Anthropometric safety measures | Over 30 days
  Blood pressure, Heart Rate, Weight, BMI
Safety and Tolerability: Number of Adverse Events | Over 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada